CLINICAL TRIAL: NCT00971334
Title: Noninvasive Screening for Fetal Aneuploidy: A New Maternal Plasma Marker
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-T21-202
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Pregnancy; Aneuploidy; Down Syndrome; Edwards Syndrome
Keywords: Down Syndrome; Aneuploidy; Amniocentesis; CVS
MeSH Terms: conditions — Aneuploidy; Down Syndrome; Trisomy 18 Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and PBMCs
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect samples for the purpose of developing a prenatal aneuploid test using circulating cell free fetal (ccff) nucleic acid from blood samples from pregnant women who have a high-risk pregnancy undergoing invasive prenatal diagnosis by chorionic villus sampling (CVS) and/or genetic amniocentesis. The results of the ccff aneuploid test will be compared to the chromosomal analysis obtained via CVS or amniocentesis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female
* Subject is pregnant
* Subject is 18 years of age or older
* Subject provides a signed and dated informed consent
* Subject agrees to provide a 30-50mL blood sample
* Subject is at increased risk for Down syndrome or other aneuploidies (greater than or equal to 35 years of age at time of delivery, elevated risk by maternal serum markers including Triple, Quad and integrated test, fetal birth defects or markers identified by ultrasound or family history of aneuploidy).
* Subject plans to undergo an amniocentesis and/or CVS procedure
* Subject agrees that the FISH, karyotype, and/or QF-PCR results obtained via the invasive procedure will be provided

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are scheduled to undergo a CVS or amniocentesis procedure and will receive the FISH, karyotype and/or QF-PCR results from the procedure.
Sampling Method: Probability Sample
Enrollment: 2502 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan T Bombard, MD, Study Director — Sequenom, Inc.
Locations (35):
- United States (30):
  - University of South Alabama, Mobile, Alabama
  - Grossmont Center for Clinical Research, La Mesa, California
  - IGO, San Diego, California
  - San Diego Perinatal Center, San Diego, California
  - Women's Healthcare at Frost Street, San Diego, California
  - Poway Womens Care, San Diego, California
  - Visions Clinical Research, Boynton Beach, Florida
  - University of Miami, Miami, Florida
  - South Florida Perinatal Medicine, Miami, Florida
  - Global Ob/Gyn Centers, Pembroke Pines, Florida
  - Discovery Clinical Research, Sunrise, Florida
  - Sheridan Clinical Research, Sunrise, Florida
  - Fetal Diagnostic Institution of the Pacific, Honolulu, Hawaii
  - Women's Clinic, Boise, Idaho
  - Reproductive Genetics Institute, Chicago, Illinois
  - Spectrum Health - Maternal Fetal Medicine, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St Louis University, St Louis, Missouri
  - Methodist Hospital, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Complete Healthcare for Women, Columbus, Ohio
  - Clinical Trials of America, Eugene, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Kingsport Perinatology, Kingsport, Tennessee
  - Perinatal Research Center, Nashville, Tennessee
  - Tenessee Maternal Fetal Medicine, Nashville, Tennessee
  - Houston Perinatal Associates, Houston, Texas
- France (5):
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hopital Cochin Port Royal, Paris
  - Hopital Robert Debre, Paris
  - Hopital Paule de Viguier - CHU Toulouse, Toulouse
  - Centre Hospitalier Regional et Universitaire - Hopital Bretonneau, Tours